CLINICAL TRIAL: NCT01986998
Title: Multicenter, Randomized, Double-blind Clinical Trial to Compare the Clinical and Radiological Efficacy of 625 mg Versus 1250 mg of Oral Methylprednisolone in Patients With Multiple Sclerosis in Relapse.
Brief Title: Study to Compare the Clinical and Radiological Efficacy of 625 mg Versus 1250 mg of Oral Methylprednisolone in Patients With Multiple Sclerosis in Relapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Cristina Ramo, Cristina Ramo, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: oral-CORTEM; 2012-001965-34 (EudraCT Number)
Record Dates: First submitted 2013-01-11; First posted 2013-11-19 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis relapse; oral methylprednisolone; EDSS; gadolinium
MeSH Terms: conditions — Multiple Sclerosis | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oMP 1250 mg: Group A (Active Comparator): Methylprednisolone 1250 mg/24h x3 days
  Interventions: Drug: Methylprednisolone 1250 mg/24h x3 days
- oMP 625 mg: Group B (Active Comparator): Methylprednisolone oral 625 mg/24h x3 days
  Interventions: Drug: Oral Methylprednisolone 625 mg/24h x3 days

INTERVENTIONS:
Drug: Methylprednisolone 1250 mg/24h x3 days — Oral Methylprednisolone 1.250 mg daily, over 1 hour and during 3 consecutive days. 13 capsules will be administered (12 capsules of 100 mg and 1 capsule of 50 mg)
  Other Names: Group A
  Arms: oMP 1250 mg: Group A
Drug: Oral Methylprednisolone 625 mg/24h x3 days — Oral Methylprednisolone 625 mg daily, over 1 hour and during 3 consecutive days. 13 capsules will be administered (6 capsules of 100 mg, 1 capsule of 25 mg and 6 capsules of placebo with the same appearance of capsules of 100 mg)
  Other Names: Group B
  Arms: oMP 625 mg: Group B

SUMMARY:
The investigators plan to carry out a multicenter randomized clinical trial and MRI study of high-dose oMP (1250mg/day for 3 days) versus lower-high dose oMP (625mg/day for 3 days) and demonstrated that lower-high dose of oMP is as effective as a higher-high dose of oMP in acute relapse of multiple sclerosis (MS). If it is shown, our purpose is to promote this therapeutic regimen because it is safer for the patient (less adverse effects) and less costly to the healthcare system.

DETAILED DESCRIPTION:
DESIGN: Phase IV clinical trial, multicentre, randomized and double blind, active drug controlled and parallel groups. Patients will be randomised to a high dose of oMP vs a lower-high dose of oral Methylprednisolone (oMP).

SETTING: 9 MS Units from 9 hospitals of the public health system with extensive experience in treating patients with MS and design and participation in clinical trials.

PROCEDURES:

After signing the informed consent, the inclusion and exclusion criteria specific to the study will be checked. The diagnostic test will take place prior to administration of study medication and will include medical history, neurological examination (EDSS measurement) taking of vital signs (blood pressure, heart rate and body temperature) and MRI. Concomitant medication will be checked. Patients will be instructed about the requirements during the study.

The trial medication will be provided to the patient in the medical office (day 1 of the study), where the patient will remain until the intake. This action will be repeated the following 2 days. The latency period from the beginning of the relapse until the start of treatment will be registered. The questionnaires of tolerance will be completed.

Day 1 will be defined as the first day on which first dose of oMP is administered.

Once given the treatment under study, the adverse events reported spontaneously or after question will be collected.

There will be follow-up visits at 7 and 28 days, and 3 months after initiation of treatment. At baseline, prior to drug administration, and on days 7 and 28 after initiation of treatment, a brain MRI with and without contrast will be performed. In case of adverse events or laboratory abnormalities, the patients could have an accessory follow-up visits until resolution.

Randomization will be performed on the day of administration (day 1)

The treatments are:

Group A: Methylprednisolone 1250 mg / day orally for 3 days Group B: Methylprednisolone 625 mg / day orally for 3 days

ELIGIBILITY:
Inclusion Criteria:

1. Relapsing-remitting MS (Mc Donald criteria 2010) regardless being under immunomodulatory treatment
2. EDSS (previous to relapse) between 0 and 5
3. MS relapse of moderate intensity (EDSS increase from 1 to 2.5 points) or severe intensity (EDSS increase > 3 points)

   * If EDSS previous relapse is available:

     * optic neuritis, myelitis or brainstem relapse: the EDSS should increase of 1 point in visual, pyramidal or brainstem system function
     * relapse in other location or uncertain location: the EDSS should increase at least 1 point
   * If EDSS previous relapse is not available:

     * optic neuritis, myelitis or brainstem relapse: the visual, pyramidal or brainstem system function should be > 2 points.
     * relapse in other location or uncertain location: EDSS should be > 2 points
4. Recent clinical relapse onset (<15 days) without fever
5. One month of clinical stability prior to relapse
6. Signed informed consent
7. Capacity to ingest the medication.

Exclusion Criteria:

1. Doubts about the diagnosis of multiple sclerosis
2. First episode of inflammatory neurological disease
3. Secondary progressive MS or primary progressive MS
4. Symptoms with lasted less than 24 hours of evolution
5. Any degree of subjective or objective remission
6. Treatment with corticosteroids during the previous 30 days
7. Patients with immunosuppressive treatment (azathioprine, mitoxantrone, cyclophosphamide) or Natalizumab or Fingolimod
8. Pregnancy or breastfeeding women or women of childbearing potential not using contraceptive measures
9. Diseases with a contraindication of treatment with corticosteroids
10. History of serious adverse reaction or hypersensitivity to drugs related to study medication
11. Patients who could not be regular MRI, not collaborators or who requires anesthesia.
12. Lactose intolerance
13. Patients with allergies to contrast used in MRI
14. Patients with renal impairment

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Disability scale of Kurtzke EDSS score | up to day 91

SECONDARY OUTCOMES:
Adverse events / tolerability | Baseline and day 29
Disability scale of Kurtzke EDSS score | Baseline and day 8
The number and volume of active lesions (measured by the T2 or gadolinium enhancement), the number of new active lesions and the percentage of active lesions at baseline that becomes black holes | day -1 and day 29
Adverse events / tolerability | Baseline and day 8
Questionnaire MSQOL-54 | Baseline and day 8
Questionnaire MSQOL-54 | Baseline and day 29

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ramo, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (8):
- Spain (8):
  - Hospital Universitari Germans Trias I Pujol de, Badalona, Barcelona
  - Hospital Del Mar, Barcelona, Barcelona
  - Hospital de Mataró, Barcelona, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Barcelona
  - Hospital de Sant Joan Despí Moisés Broggi, Barcelona, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona, Girona
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida, Lleida
  - Hospital de Sant Pau I Santa Tecla, Tarragona, Tarragona

REFERENCES:
- [Derived] Hervas-Garcia JV, Ramio-Torrenta L, Brieva-Ruiz L, Batlle-Nadal J, Moral E, Blanco Y, Cano-Orgaz A, Presas-Rodriguez S, Torres F, Capellades J, Ramo-Tello C. Comparison of two high doses of oral methylprednisolone for multiple sclerosis relapses: a pilot, multicentre, randomized, double-blind, non-inferiority trial. Eur J Neurol. 2019 Mar;26(3):525-532. doi: 10.1111/ene.13851. Epub 2018 Nov 16. PMID 30351511